CLINICAL TRIAL: NCT01269684
Title: A 6-Month Open Pilot Study to Investigate the Safety and Tolerability of Immediate Conversion From Calcineurin Inhibitor Tacrolimus to Everolimus in Stable Maintenance Renal Transplant Recipients
Brief Title: Immediate Conversion From Tacrolimus to Everolimus in Stable Maintenance Renal Transplant Recipients
Acronym: HERMES
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: No patient has never been included in the trial
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001ACH04
Record Dates: First submitted 2010-10-05; First posted 2011-01-04 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Kidney Transplantation
Keywords: Kidney; renal; transplantation; tacrolimus; everolimus; stable allograft recipients
MeSH Terms: interventions — Everolimus

ARMS (1):
- 1 (Experimental): Initial dose 1.5 mg b.i.d. Target blood trough level 4-10 ng/ml
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — Initial dose 1.5 mg b.i.d. Target blood trough level 4-10 ng/ml
  Other Names: Certican

SUMMARY:
The purpose of this study is to investigate safety and tolerability of an immediate conversion from Tacrolimus to everolimus in stable renal allograft recipients.

Interest in developing CNI-free regimens using other agents such as the proliferation signal inhibitor everolimus.

ELIGIBILITY:
Inclusion criteria

* Primary or secondary renal transplantation in the past 12-36 months.
* Current immunosuppressive therapy consisting of Tacrolimus together with MMF +/-corticosteroids.
* Moderately impaired renal function

Exclusion criteria

* Multi-organ recipients or previous transplantation with an organ other than a kidney.
* Acute rejection episodes in the last 6 months.

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-08 (Actual); Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Routine safety laboratory | At baseline
Routine safety laboratory | Week 1
Routine safety laboratory | Month 1
Routine safety laboratory | Week 2
Routine safety laboratory | Week 3
Routine safety laboratory | Month 2
Routine safety laboratory | Month 4
Routine safety laboratory | Month 6

SECONDARY OUTCOMES:
renal function | At baseline
renal function | Weeks 1, 2 and 3
renal function | Months 1, 2, 4 and 6

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Zurich, Switzerland